CLINICAL TRIAL: NCT06610656
Title: The Effect of White Noise and Pacifier Applications on Pain and Crying Time in Newborns in the Postoperative Period
Brief Title: White Noise and Pacifier Use on Postoperative Pain and Crying in Newborns
Acronym: CLİNİCAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Arzu Bahar, Associate Pofessor, Yuksek Ihtisas University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ABAHAR-004
Record Dates: First submitted 2024-09-16; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Pain
Keywords: white noise; pacifier; newborn; surgery
MeSH Terms: conditions — Pain | interventions — Pacifiers

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment design in which participants are assigned to one of two intervention groups. Group 1 will receive pacifier and white noise therapy, while Group 2 will receive pacifier therapy only. Each group will be treated independently, and there will be no crossover between the groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: n this study, both participants and investigators are masked to the group assignment. Participants will not be aware of whether they are receiving pacifier therapy alone or in combination with white noise therapy. Investigators will not know the specific group assignments during the intervention to minimize bias in observations and assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- White noise and pacifier applications group (Experimental): In this group, infants will receive pacifier and white noise therapy. The white noise will be used to enhance the quality of sleep and reduce restlessness in infants. During the intervention, participants will receive pacifiers, and white noise will be continuously administered.
  Interventions: Other: Pacifier and White Noise Therapy
- pacifier applications group (Active Comparator): In this group, infants will receive only pacifier therapy. The aim is to provide comfort and support for sleep through the use of pacifiers. White noise will not be utilized in this group. This intervention focuses solely on assessing the effects of pacifier use without any additional auditory stimuli
  Interventions: Other: pacifier therapy

INTERVENTIONS:
Other: Pacifier and White Noise Therapy — Infants will receive both pacifier and white noise therapy to enhance sleep quality and reduce restlessness
  Arms: White noise and pacifier applications group
Other: pacifier therapy — Infants will receive pacifier therapy to enhance sleep quality and reduce restlessness
  Arms: pacifier applications group

SUMMARY:
The study was conducted to determine the effect of white noise and pacifier applications on pain and crying time during painful interventions in newborns who underwent surgery

DETAILED DESCRIPTION:
Newborns most often experience painful procedures such as heel blood collection and peripheral venous catheter placement in the neonatal intensive care unit. Exposure to pain early in life has even been shown to increase the risk of developing problems (chronic pain, anxiety, and depressive disorders) in adulthood. This result implies that newborn or child pain should be adequately managed. Thus, pain in newborns or children should be prevented before it occurs, and if it cannot be prevented, it should be determined in the early period and the pain should be alleviated. Managing this pain in newborns should be one of the primary duties of newborn nurses. The first and most important determinant in relieving pain is determining the severity of pain, and non-pharmacological or pharmacological methods should be preferred according to the severity of the pain. Many non-pharmacological methods are used to manage pain that may occur in interventional procedures. Some of these methods are: giving sugar solution, kangaroo care, positioning (Kaşıkçıoğlu, 2014), breast milk and breastfeeding and swaddling, listening to music, lullaby. Two other effective methods are non-nutritive suction and white noise. As a result of studies, it was proven that the use of multiple non-pharmacological methods together was much more effective in reducing pain. Within the scope of the research, no research was found in the literature regarding which application - white noise or pacifier - could be more effective. By examining this information, the effects of the two effective methods on pain management and crying time in newborns in the postoperative period were examined in this study.

ELIGIBILITY:
Inclusion Criteria:

* Birth weight over 1500 grams

  * Having passed the newborn hearing screening test
  * Having a history of previous surgery (excluding brain surgeries)
  * Not using sedative substances (dormicum, fentanyl)
  * Not using opioids
  * Having a full stomach 30 minutes before painful interventions
  * Having permission from their mothers
  * Newborns undergoing blood transfusion only

Exclusion Criteria:

* Being intubated

  * Having hiberbilirubinemia
  * Birth weight below 1500 grams
  * Having cerebral palsy
  * Having hydrocephalus
  * Having spina bifida
  * Having had brain surgery

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
1. Neonatal Pain Scale (NIPS | 20 minutes
  The factors evaluated in the newborn baby pain scale are facial expression, arms, legs, oxygen saturation, arousal, breathing pattern, crying, heart rate. It can be preferred in post-operative pain. It can be used in procedural pain. It has a total of 8 parameters. The highest score can be given is 7. 0 points = no pain, 1-2 points = mild pain, 3-4 points = moderate pain, >4 points = severe pain is accepted.

CONTACTS AND LOCATIONS:
Overall Officials: arzu bahar, Principal Investigator — Yüksek Ihtisas University
Locations (1):
- Yüksek Ihtisas Üniversity, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No